CLINICAL TRIAL: NCT07352202
Title: Evaluation of Gastric Emptying and Residual Volume Using Ultrasound in Mechanically Ventilated Intensive Care Patients Receiving Different Enteral Nutrition Solutions
Brief Title: Ultrasound Assessment of Gastric Emptying in Mechanically Ventilated ICU Patients
Acronym: GASTRIC-USG
Status: Recruiting | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-395
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gastric Ultrasound
Keywords: gastric ultrasound; ıntensive care unit; gastric residual volume
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard Enteral Nutrition: Mechanically ventilated intensive care unit patients receiving standard enteral nutrition as part of routine clinical care.
  Interventions: Other: Enteral Nutrition (Routine Clinical Care)
- Specialized Enteral Nutrition: Mechanically ventilated intensive care unit patients receiving specialized enteral nutrition formulations according to routine clinical practice.
  Interventions: Other: Enteral Nutrition (Routine Clinical Care)
- Water Administration: Mechanically ventilated intensive care unit patients receiving water administration via nasogastric tube as part of routine care.
  Interventions: Other: Enteral Nutrition (Routine Clinical Care)

INTERVENTIONS:
Other: Enteral Nutrition (Routine Clinical Care) — Enteral nutrition administered according to routine clinical practice without protocol-driven assignment or modification.

SUMMARY:
This prospective observational study aims to evaluate dynamic changes in gastric volume and gastric emptying time using bedside gastric ultrasound in mechanically ventilated intensive care unit patients. The study compares gastric emptying patterns among patients receiving different types of enteral nutrition solutions as part of routine clinical care.

DETAILED DESCRIPTION:
This prospective observational study is designed to evaluate gastric emptying and changes in gastric volume using bedside gastric ultrasound in mechanically ventilated intensive care unit patients. Ultrasound examinations will be performed at predefined time points to assess gastric residual volume and gastric emptying patterns.

Patients receiving different types of enteral nutrition solutions as part of routine clinical care will be evaluated and compared. Gastric measurements will be obtained using standardized ultrasound techniques by trained clinicians.

The study aims to identify differences in gastric emptying dynamics associated with various enteral nutrition formulations and to assess the feasibility of bedside ultrasound as a non-invasive tool for monitoring gastric function in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Mechanically ventilated patients admitted to the intensive care unit
* Presence of a nasogastric tube
* Hemodynamically stable patients receiving enteral nutrition as part of routine clinical care

Exclusion Criteria:

* Recent abdominal surgery within the first 24 hours
* Major abdominal trauma or burns
* Significant ascites
* Inadequate ultrasound window (e.g., severe meteorism)
* Hemodynamic instability
* Contraindication to enteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who are mechanically ventilated and admitted to the intensive care unit. Eligible patients are those receiving enteral nutrition via a nasogastric tube as part of routine clinical care and who are hemodynamically stable. Patients will be observed prospectively without any protocol-driven intervention.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Change in Gastric Volume Estimated by Ultrasound | Baseline and up to 60 minutes after enteral feeding
  Dynamic changes in gastric volume estimated using ultrasound-derived antral cross-sectional area measurements at predefined time points before and after enteral feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Berfin Gizem G Özelsel, MD, Principal Investigator — Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Locations (1):
- Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional data protection policies and the inclusion of critically ill patients. Data will be analyzed and reported in an aggregated and anonymized manner.